CLINICAL TRIAL: NCT03958019
Title: Rehabilitation Strategies Following Oesophagogastric and Hepatopancreaticobiliary Cancer (RESTORE II) - A Randomised Controlled Trial
Brief Title: Rehabilitation Strategies Following Oesophagogastric and Hepatopancreaticobiliary Cancer
Acronym: RESTORE II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other); St. James's Hospital, Ireland (Other); St Vincent's University Hospital, Ireland (Other); Tallaght University Hospital (Other)
Responsible Party: Principal Investigator, Prof Juliette Hussey, Professor Juliette Hussey, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRB-DIFA RESTORE II Trial
Record Dates: First submitted 2019-04-02; First posted 2019-05-21 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Oesophageal Cancer; Gastric Cancer; Liver Cancer; Pancreatic Cancer
Keywords: Rehabilitation; Exercise; Diet; Education; Survivor-ship
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Convergent parallel mixed methods design
Who Masked: Outcomes Assessor
Masking Description: Study outcomes will be assessed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 12 week multidisciplinary program consisting of; i) supervised and home-based aerobic and resistance training, ii) 1:1 dietary counselling, and iii) group education sessions.
  Interventions: Other: RESTORE II Program
- Control (No Intervention): Usual care control group

INTERVENTIONS:
Other: RESTORE II Program — Detailed in arm description
  Arms: Intervention Group

SUMMARY:
The RESTORE II randomized controlled trial will examine the efficacy of a 12 week multidisciplinary rehabilitation program consisting of supervised and home-based exercise,1:1 dietetic counselling, and group education sessions for survivors of upper gastrointestinal cancer, namely cancers of the oesophagus, stomach, pancreas, and liver.

DETAILED DESCRIPTION:
Curative treatment for upper gastrointestinal (UGI) cancers is associated with numerous side-effects including sarcopenia and nutritional compromise, increasing morbidity, compromising functional capacity and decreasing health-related quality of life (HR-QOL) in survivorship. As survival improves in UGI cancer, there is increasing focus on optimizing survivorship, however research examining rehabilitation programs in this newly-emergent complex clinical cohort is lacking.

The investigators recently designed, implemented, and evaluated the Rehabilitation Strategies following Oesophagogastric Cancer (RESTORE) program, a novel multidisciplinary rehabilitation program tailored for oesophagogastric cancer survivorship. The feasibility and preliminary efficacy of the RESTORE program was established and there is now recognized need to further examine program efficacy in a definitive trial.

Using a convergent parallel mixed-methods design, RESTORE II, implemented as a 2-armed randomized controlled trial, will examine if multidisciplinary rehabilitation can improve functional capacity and HRQOL in UGI cancer survivors. RESTORE II will prescribe a 12-week program of supervised aerobic and resistance training, self-directed unsupervised exercise, individualized dietetic counselling and multidisciplinary education for patients who are >3 months following oesophagectomy, gastrectomy, pancreaticoduodenectomy, or major liver resection. A sample of 60 participants per arm will be recruited to establish a mean increase in functional capacity (cardio-respiratory fitness) of 3.5 ml/kg/min with 90% power, 5% significance and 20% drop-out.

Quantitative assessments including cardiopulmonary fitness and functional exercise capacity will be completed at baseline, post-intervention and 3-months post-intervention (Objective 1). HR-QOL will be quantitatively assessed pre and post-intervention, at 3-months post-intervention and 1 year post-enrollment (Objective 2). Impact on physical, mental and social well-being will be qualitatively examined during focus groups immediately post-intervention and 3-months post-intervention (Objective 3). The implementation costs of RESTORE II will be analysed in consideration of clinician salaries, overheads and equipment costs (Objective 4). Bio-samples will be collected pre and post-intervention and 3-months post-intervention, establishing the first National UGI Cancer Survivorship Biobank (Objective 5). A patient centered approach to enhancing trial recruitment in this complex cohort will also be evaluated (Objective 6).

Following this evaluation, the RESTORE II program will provide a unique model of multidisciplinary rehabilitation in nutritionally complex UGI cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients >3-months post oesophagectomy, total gastrectomy, pancreaticoduodenectomy or major liver resection +/- neo-adjuvant/adjuvant chemo/chemoradiotherapy with curative intent
* Completion of adjuvant oncological therapy
* Successful completion of baseline cardiopulmonary exercise test
* Medical clearance to participate.

Exclusion Criteria:

* Ongoing serious post-operative morbidity
* Evidence of active or recurrent disease
* Co-morbidities that would preclude safe exercise participation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness from Baseline | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Cardiorespiratory fitness will be determined by Cardiopulmonary Exercise Test (CPET)

SECONDARY OUTCOMES:
Physical Performance | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Physical Performance will be measured with the Short Physical Performance Battery (SPPB)
Lower Limb Muscle Strength | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Lower limb muscle strength (llbs)will be measured by a leg press 1-RM
Hand Grip Strength | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Hand grip strength (kg) will be measured with hand held dynamometry
Physical Activity | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Physical Activity levels will be measured by accelerometry (ACTIGRAPH GT3X+)
Body Mass Index | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Body mass index will be measured as the ratio of weight (kg) to height in metres squared.
Waist Circumference | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Waist circumference (cm) will be measured at the mid-point between the iliac crest and the 12th rib following gentle expiration.
Mid Arm Circumference | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Mid Arm circumference (cm) will be measured at the mid-point between the olecranon process of the ulna and the acromion process of the scapula.
Fat Mass | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Fat mass(kg) will be measured with the Seca mBCA 515.
Fat Free Mass | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Fat free mass (kg) will be measured with the Seca mBCA 515.
Skeletal Muscle Mass | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Skeletal muscle mass(kg) will be measured with the Seca mBCA 515.
Dietary Quality | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Dietary quality will be scored using the WCRF/AICR index which determines adherence to healthy eating guidelines for cancer survivors.
Health Related Quality of Life | Baseline (T0), Immediately after the program intervention (T1), Three month Follow-up (T2), One-year post intervention (T3)
  Quality of Life will be determined by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30).
  Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Health Related Quality of Life (Specific to Oesophago-gastric cancer) | Baseline (T0), Immediately after the program intervention (T1), Three month Follow-up (T2), One-year post intervention (T3)
  For Oesophago-gastric Cancer Patients Quality of Life will be further assessed with the European Organisation for Research and Treatment of Cancer Oesophago-gastric Cancer Subscale the QLQ-OG25.
  Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Health Related Quality of Life (Specific to Hepatocellular carcinoma) | Baseline (T0), Immediately after the program intervention (T1), Three month Follow-up (T2), One-year post intervention (T3)
  For Liver Cancer Patients Quality of Life will be further assessed with the European Organisation for Research and Treatment of Cancer Core Hepatocellular carcinoma subscale (QLQ-HCC18) Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Health Related Quality of Life (Specific to Pancreatic carcinoma) | Baseline (T0), Immediately after the program intervention (T1), Three month Follow-up (T2), One-year post intervention (T3)
  For Pancreatic Cancer Patients Quality of Life will be further assessed with the European Organisation for Research and Treatment of Cancer Pancreatic cancer Subscale (QLQ-PAN26).
  Scores are reported on a linear scale from 0-100. A high score on a functional scale indicates greater function. A high score on a symptom scale indicates greater symptom burden.
Fatigue | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Fatigue will be assessed using the Multidimensional Fatigue Inventory (MFI-20) questionnaire. It is scored from 0-20. A cut off score of >or =13 indicates severe fatigue.
Qualitative Approach | Immediately after the program intervention and Three-months post intervention
  Focus groups and interviews will be carried out with participants from the intervention arm to gain their perspectives of the impact of the program on physical and mental well-being.
Cost Analysis | Up to 1 year post program completion
  The costs of the program will be set against the effects on HRQOL
Bio-sample Collection | Baseline (T0), Immediately after the program intervention (T1), and Three month Follow-up (T2)
  Serum and Plasma samples will be collected at each time-point to establish a survivorship Biobank for UGI cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Hussey, PhD, Principal Investigator — Professor in Physiotherapy
Locations (1):
- Trinity College, Dublin, Leinster, Ireland

REFERENCES:
- [Derived] O'Neill L, Knapp P, Doyle SL, Begic S, Smyth E, Kearney N, Grehan S, Parker A, Browne P, Segurado R, Connolly D, O'Sullivan J, Reynolds JV, Guinan E, Hussey J. Can a Public and Patient Involvement (PPI) Informed Participant Information Leaflet (PIL) Improve Trial Recruitment, Retention, and Quality of Decision Making? Results of a Randomised Controlled Double-Blind Study Within a Trial (SWAT). Health Expect. 2025 Jun;28(3):e70321. doi: 10.1111/hex.70321. PMID 40485109
- [Derived] O'Neill L, Murphy F, Reidy D, Poisson C, Hussey J, Guinan E. Development and Initial Implementation of a Clinical Monitoring Strategy in a Non-regulated Trial: a research note from the ReStOre II Trial. HRB Open Res. 2024 Oct 18;6:46. doi: 10.12688/hrbopenres.13763.3. eCollection 2023. PMID 39280895
- [Derived] O'Neill L, Knapp P, Doyle SL, Guinan E, Parker A, Segurado R, Connolly D, O'Sullivan J, Reynolds JV, Hussey J. Patient and family co-developed participant information to improve recruitment rates, retention, and patient understanding in the Rehabilitation Strategies Following Oesophago-gastric and Hepatopancreaticobiliary Cancer (ReStOre II) trial: Protocol for a study within a trial (SWAT). HRB Open Res. 2020 Nov 10;2:27. doi: 10.12688/hrbopenres.12950.2. eCollection 2019. PMID 33392438
- [Derived] O'Neill L, Guinan E, Doyle S, Connolly D, O'Sullivan J, Bennett A, Sheill G, Segurado R, Knapp P, Fairman C, Normand C, Geoghegan J, Conlon K, Reynolds JV, Hussey J. Rehabilitation strategies following oesophagogastric and Hepatopancreaticobiliary cancer (ReStOre II): a protocol for a randomized controlled trial. BMC Cancer. 2020 May 13;20(1):415. doi: 10.1186/s12885-020-06889-z. PMID 32404096